CLINICAL TRIAL: NCT01482130
Title: Preventing Osteoporosis: The Effect of High Intensity Strength Training on Bone Mineral Density in Young and Healthy Women
Brief Title: High Intensity Strength Training & Bone Mineral Density in Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REK-2011/2039
Record Dates: First submitted 2011-11-16; First posted 2011-11-30 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Osteoporosis
Keywords: Exercise; osteoporosis; prevention
MeSH Terms: conditions — Osteoporosis; Motor Activity | interventions — Health Planning Guidelines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training group (Experimental): All participants in the training group will pursue a 12 weeks of strength training.
  Interventions: Behavioral: Heavy, explosive strength training
- Controls (Other): The control group will be encouraged to follow a training program according to recommended exercise guidelines
  Interventions: Behavioral: recommendations

INTERVENTIONS:
Behavioral: Heavy, explosive strength training — All participants of the training group will pursue a 12 weeks of heavy, explosive strength training, 3 sessions a week for a total of 36 sessions. The training session will include one squat exercise only, which allows muscle contraction of the quadriceps from a 90° bend at the knees to straight legs.
  Arms: Training group
Behavioral: recommendations — The control group will be encouraged to follow a training program according to recommended exercise guidelines:
  * Weight bearing activities (walking, jogging or strength training)
  * 30 - 60 minutes, 3 - 5 times each week
  * A total of 2 - 3 hours each week should be achieved
  Arms: Controls

SUMMARY:
The current guidelines emphasize the prevention of bone loss, by building up bone mass in young age, as one of the most important measures to reduce the incidence of osteoporosis. Strength training and "explosive" exercises have been shown to have beneficial effects on bone mass and bone metabolism in both young and postmenopausal women. However, meta-analysis concludes that it is still unclear what type of exercises, intensity and execution that is most effective for skeletal adaptations. The following study will examine the effect of 12 weeks of heavy, explosive strength training on bone mineral density and bone metabolism in young, healthy girls aged 18-30 years.

DETAILED DESCRIPTION:
Background:

Osteoporosis is a progressive, systemic skeletal disorder characterized by low bone mineral density (BMD), and deterioration of the microarchitecture of bone tissue, with a consequent increase in bone fragility and susceptibility to fracture. Typically the disease shows no symptoms until a fracture occurs, hence referred to as the "silent epidemic". In Norway one of two women and one of four men experience a fragility fracture after the age of 50. The loss of bone strength with age likely reflects the skeletal response to hormonal changes and the mechanical environment with decreased physical activity. Osteoporotic fractures often happen as a consequence of minimal injury, especially at the hip, spine and wrist. Hip fracture is associated with excess mortality during the first year after fracture ranging from 8.4% to 36%. The increased mortality risk may persist for several years thereafter, highlighting the need for interventions to reduce this risk. Osteoporosis is a common disease and recognized as a global problem by the WHO.

The American College of Sport Medicine suggests exercise as a countermeasure against bone loss in postmenopausal woman and elderly subjects. Peak bone mass is thought to be attained by the end of the third decade, hence the early adult years might be the final opportunity for its augmentation. It is indicated that optimizing peak bone mass may have long-term effect on bone health. Intervention studies with young women show that high impact exercises may improve BMD in young adults. High intensity strength training also seems to effectively improve BMD and the ratio of bone turnover markers. Furthermore, an explosive execution of movement may be important for obtaining BMD improvements from resistance training. Maximal strength training (MST) is characterized by high mobilization of force, high loads, and few repetitions (3-5 reps.) per set with emphasis on maximal force mobilization in the concentric part of the movement. Recent studies have shown that MST is highly efficient for improving maximal strength (1RM) and rate of force development (RFD). Parameters such as 1RM and RFD are closely related to BMD. In addition, a recent study from our group showed that 12 weeks of MST training (three times each week) improved bone mass in the hip and spine of postmenopausal women, diagnosed with osteoporosis (article in preparation). In the present study we want to investigate the impact of heavy, explosive strength training on bone mass and bone metabolism in young and healthy woman which have not yet reached peak bone mass.

Physical activity and BMD:

One of the main factors responsible for the high incidence of osteoporosis is physical inactivity. Several studies have shown that physical activity can lead to an increase in BMD. Resistance- and impact exercises have shown to be most effective. A number of studies performed with sedentary young women performing high impact training has shown significant improvement in BMD at the femoral neck and lumbar spine. A study with postmenopausal women showed that power training is more effective in maintaining BMD in the lumbar spine and total hip than conventional strength training.

The effect of training at the cellular and tissue level can be divided into 3 main factors:

* Increased osteoblast activity and bone formation
* Reduced osteoclast activity and bone resorption
* Increased stability of the bone's architectural structure

In terms of prevention of osteoporosis the current exercise guidelines, according to the WHO, is encouragement of a physically active lifestyle. Weight bearing activities, preferably resistance training are recommended for patients with osteoporosis. Peak bone mass is an important factor in determining long-term fracture risk. Therefore, effective strategies to maximize peak bone mass in young adults are essential. Evidence indicates that resistance and high-impact exercise are the most beneficial to maintain and optimize peak bone mass in young adults. However, studies investigating such exercises are not altogether conclusive, and the mode of exercise, regarding type of exercise, intensity and execution, still remains unclear. Since MST exercise may increase bone mass in osteoporotic women, and improves 1RM and RFD (which are closely related to skeletal health) we wish to investigate the potential of MST training to increase bone mass and improve bone metabolism in young female adults, who have not yet reached peak bone mass.

Goals of the study:

1. Investigate the effect of heavy, explosive strength training on bone mineral density compared to a control group in young, healthy women over a period of 3 months.
2. Study the effect of this training intervention on bone formation and resorption markers
3. Study the effect on physical capacity measurements.

ELIGIBILITY:
Inclusion Criteria:

* Participants include young and healthy women between the ages of 18-30, who have not engaged in strength training for the last 6 months.

Exclusion Criteria:

* Subjects will be excluded from the study if they have any condition that preclude them from taking part in the exercise testing procedures or the 24 week exercise program or if they fail to obtain the required amount of training sessions.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Baseline and 12 weeks
  (Dual X-ray Absorptiometry)

SECONDARY OUTCOMES:
Serum markers of bone metabolism | Baseline and 12 weeks
  Blood samples will be drawn for analyses of bone metabolism and markers of bone formation; osteoprotegerin (OPG) and Type I procollagen N-terminal propeptide (PINP). Furthermore, Type 1 collagen C-breakdown products (CTX) and receptor activator of NF kappa B ligand (RANKL) which are the key regulators of bone resorption, will be analyzed at the start and end of the study.
Body composition | Baseline and 12 weeks
  Lean- versus fat mass, measured by Dual X-ray Absorptiometry (DXA).
Maximal muscle strength | Baseline and 12 weeks
  Measured as one repetition maximum in a squat exercise machine.
Rate of force development | Baseline and 12 weeks
  Maesured dynamic in a squat exercise maschine, and isometric at 90 degree angle in the knee joint.

CONTACTS AND LOCATIONS:
Overall Officials: Unni Syversen, MD, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Sor.tronderlag, Norway

REFERENCES:
- [Result] Mosti MP, Carlsen T, Aas E, Hoff J, Stunes AK, Syversen U. Maximal strength training improves bone mineral density and neuromuscular performance in young adult women. J Strength Cond Res. 2014 Oct;28(10):2935-45. doi: 10.1519/JSC.0000000000000493. PMID 24736773